CLINICAL TRIAL: NCT06961409
Title: Evaluation of Salivary Granulocyte-Macrophage Colony-Stimulating Factor, Macrophage Inflammatory Protein and Interleukin-1β Levels in Individuals With Different Periodontal Conditions
Brief Title: Assessment of Salivary GM-CSF, MIP, and IL-1β Levels in Subjects With Varying Periodontal Conditions
Status: Recruiting | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Mehmet Sait Bilgic, Research Assistant, Izmir Katip Celebi University
Other Study IDs: 2024--SAEK-0039
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Periodontal Diseases; Periodontitis; Gingivitis; Periodontal Health
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Unstimulated whole saliva samples collected from healthy, gingivitis, and periodontitis subjects will be retained for biomarker analysis. No DNA extraction will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Periodontium: Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: Saliva obtaining
- Gingivitis: Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: Saliva obtaining
- Periodontitis: Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: Saliva obtaining

INTERVENTIONS:
Diagnostic Test: Saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated saliva was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Tubes were stored at -80ºC until the day of analysis.
  Groups: Healthy Periodontium
Diagnostic Test: Saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated saliva was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Tubes were stored at -80ºC until the day of analysis.
  Groups: Gingivitis
Diagnostic Test: Saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated saliva was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Tubes were stored at -80ºC until the day of analysis.
  Groups: Periodontitis

SUMMARY:
In order to determine the pathogenesis of chronic inflammatory diseases, the levels of various cytokines are examined in tissues and fluids taken from the body. In recent publications, the role of Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF), Macrophage Inflammatory Protein (MIP)-1α and Interleukin (IL)-1β on chronic inflammatory diseases has been investigated. The aim of this study was to evaluate the levels of these cytokines in the saliva of healthy individuals with gingivitis and periodontitis.

All oral clinical parameters of 60 systemically healthy individuals (20 healthy, 20 with gingivitis and 20 with periodontitis) who applied to our clinic for routine periodontal control will be measured and saliva samples will be taken from the patients. GM-CSF, MIP-1α and IL-1β (biomarkers emphasizing inflammation in saliva samples) will be determined by enzyme-linked immunoassay (ELISA). Then, statistical analyses will be performed to interpret the difference in cytokine levels between the groups and the relationship between these cytokines and clinical parameters.

Possible significant differences in cytokine levels will reveal that these proteins and enzymes can be utilized as a diagnostic tool in periodontal diseases, to distinguish periodontal disease status from healthy, or as a guide for treatments.

DETAILED DESCRIPTION:
Periodontal disease is characterized by various microbial infections caused by only certain microbial species out of the many types of bacteria present in the oral cavity, with progressive destruction of the tissues supporting the tooth.

Gingivitis is an inflammation caused by substances secreted from microbial plaque accumulated in or near the gingival sulcus, in the gingival tissue surrounding the teeth, and develops due to bacterial plaque. Gingivitis, the mildest form of periodontal disease, is a common condition and can usually be easily treated with good oral hygiene. Gingivitis, as defined, is present in 50% to 90% of adults worldwide. It has been observed that untreated gingivitis lesions are often at risk of developing into periodontitis in individuals. Periodontal disease is a disorder that causes loss of attachment in the tissues surrounding the tooth and destruction of alveolar bone. Periodontitis, which is the main cause of tooth loss in adults, is a common health problem. The initial cause of periodontitis lesions is microbial dental plaque, which is organized on the teeth and contains many pathogenic bacteria. Within the microbial dental plaque, Porphyromonas gingivalis (Pg), Tannerella forsythensis (Tf) and Treponema denticola (Td) play a major role in the formation of active periodontitis lesions.

Although the presence of pathogens is necessary for the onset and progression of periodontal disease, this alone is not sufficient. The host immune response is the main driver of the pathologic process. A dysregulated host immune response or imbalance within the microbial community (dysbiosis) may lead to disruption of homeostasis in the periodontium, leading to destruction of the extracellular matrix and alveolar bone loss. In immune-inflammatory processes triggered by the interaction of host and bacteria, excessive release of proinflammatory cytokines such as IL-1, IL-6, IL-8, prostaglandin E2 (PGE2) and tumor necrosis factor-α (TNF-α) as well as endopeptidases such as matrix metalloproteinases (MMPs) have been found to cause periodontal destruction.

Inflammation in periodontitis and similar local inflammatory lesions and systemic connective tissue diseases causes an increase in biological mediators such as cytokines, prostaglandins and matrix metalloproteinases (MMPs) in the tissues involved and in the systemic circulation.

Members of the colony-stimulating factor (CSF) superfamily are involved in mammalian myelopoiesis, i.e. the formation of monocytes, macrophages, dendritic cells (DCs) and polymorphonuclear phagocytes (neutrophils and eosinophils). There are three main members of this family: Macrophage (M)-CSF (or CSF-1), Granulocyte (G)-CSF (or CSF-3) and Granulocyte-Macrophage (GM)-CSF (or CSF-2). They were first identified as growth factors capable of promoting myeloid colony formation from bone marrow precursors in vitro. In these three CSFs, the entire structure of phagocytes can potentially be controlled . GM-CSF, as its name suggests, was initially identified as a hematopoietic growth factor due to its ability to induce the differentiation of granulocytes and macrophages in vitro by inducing the proliferation and differentiation of bone marrow progenitor cells. However, it was later seen as a cytokine that acts through a specific receptor on myeloid cell populations such as monocytes/macrophages, neutrophils and eosinophils, activating/differentiating them and having a potential role in inflammation.Data from models of autoimmunity and chronic inflammation using mice lacking the GM-CSF gene or neutralizing monoclonal antibodies (mAbs) suggest that GM-CSF may be an important driver of tissue inflammation and associated pain. Examples include arthritis, EAE (Induced Experimental Autoimmune Encephalomyelitis), cardiovascular disease and lung disease. GM-CSF was one of the first cytokines detected in inflamed human synovial fluid and its biological effects outside the bone marrow vary depending on its location and concentration.

The role of this cytokine in regulating inflammation has made it attractive targets for therapeutic interventions, especially in the treatment of chronic inflammation and cancer. Many of these strategies target GM-CSF for its inflammatory properties. Understanding the cellular and molecular mechanisms by which GM-CSF exerts these diverse effects is essential for the development of better therapies for chronic inflammatory diseases. Antibodies targeting GM-CSF or its receptor GMRa are currently in early-stage clinical development for the treatment of rheumatoid arthritis and multiple sclerosis.

In a study by Zhu et al, salivary levels of GM-CSF were found to be specifically elevated in the erosive oral lichen planus group. GM-CSF has been shown to increase matrix metalloproteinase expression in monocyte-macrophages and in some cases may lead to the development of bone resorbing osteoclast precursors.

Macrophage Inflammatory Protein (MIP)-1α was first identified in 1988 as MIP-1α, an 8-kd protein pair partially purified from endotoxin-stimulated macrophages. MIP-1α is a C-C family chemokine that is a potent chemoattractant for monocytes and can be stimulated by lipopolysaccharide (LPS). It was named macrophage inflammatory protein because it induces neutrophil accumulation when injected into the footpads of mice.

MIP-1α is produced by cells during infection or inflammation. MIP-1α expression can be induced in various cell types including monocytes, macrophage cell lines, mast cell lines, Langerhans cells, fibroblasts and T lymphocytes.

MIP-1α plays an important role in the pathogenesis of various inflammatory diseases and conditions such as periodontitis, multiple myeloma, Sjögren's syndrome and rheumatoid arthritis . They fulfill various biological functions such as recruitment of inflammatory cells, wound healing, inhibition of stem cells and maintenance of effector immune response. MIP-1α promotes the orientation and movement of osteoclasts. It initiates the process of osteoclastogenesis by directly activating osteoclast cells.

In bone marrow samples from patients with Multiple Myeloma, MIP-1α/CCL3 mRNA expression is higher compared to healthy individuals. There is a strong positive correlation between bone resorption markers such as serum bone-specific alkaline phosphatase (S-BALP) and serum MIP-1α levels in patients with multiple lytic bone lesions.

MIP-1α has recently been shown to play a role in the regulation of tumor metastasis.

Oral squamous cell carcinoma (OSCC) patients with metastatic lymph nodes had increased MIP-1α mRNA expression compared to those with non-metastatic lymph nodes. This suggests a possible role of MIP-1α in tumor migration.

In a study conducted by Petkovic et al. in which peri-implant groove fluid was evaluated, MIP-1α values were found to be higher in peri-implant mucositis groups compared to healthy control group patients. In the same study, the mean peri-implant groove fluid values of MIP-1α were found to be statistically significantly higher in the group with advanced mucositis compared to the group with early mucositis.

IL-1, the first interleukin identified, has many biological activities. In fact, before the molecular identification of IL-1 in the mid-1980s, various biological functions of this cytokine had been studied for many years under different names such as leukocyte endogenous mediator, hematopoietin 1, endogenous pyrogen, catabolin and osteoclast activating factor. In the last decade, other members of the IL-1 family have been identified and their important roles in innate and adaptive immune responses have been established.

Many aspects of the diverse biological roles of IL-1α and its functional homolog but structurally distinct relative IL-1β have been elucidated by the Dinarello laboratory. IL-1α and IL-1β are key members of the IL-1 family, which currently consists of eleven members. IL-1α and IL-1β are key proinflammatory cytokines that exert pleiotrophic effects in various cells and play critical roles in both acute and chronic inflammatory and autoimmune disorders. These cytokines interact with two types of receptors, IL-1 type 1 receptor (IL-1RI) and IL-1 type 2 receptor (IL-1 RII).

IL-1α and IL-1β carry out signal transduction through IL-1RI. IL-1β has important homeostatic functions in the normal organism such as regulation of nutrition, sleep and temperature. However, overproduction of IL-1β is involved in pathophysiological changes that occur in different disease states such as rheumatoid arthritis, neuropathic pain, inflammatory bowel disease, osteoarthritis, vascular disease, multiple sclerosis and Alzheimer's disease. IL-1β can be released from immune cells such as keratinocytes, fibroblasts, synoviocytes, endothelial, neuronal, macrophages and mast cells and glial cells such as Schwann cells, microglia and astrocytes.

IL-1β plays a key role in the regulation of the innate immune response and underlies autoinflammatory diseases such as cryopyrin-associated periodic syndromes (CAPS) and familial Mediterranean fever (FMF).

In a study by Fonseca et al. in which peri-implant groove fluid was evaluated, the IL-1β value in peri-implant groove fluid of peri-implantitis regions was higher than that of peri-implant mucositis regions. Curtis et al. showed that IL-1β measurement can make an important contribution to clinical findings in the diagnosis of peri-implantitis.

Relvas et al. observed that salivary IL-1β levels were higher in periodontitis stage III/IV patients than in periodontally healthy control patients and periodontitis stage I/II patients. In addition, IL-1β was found to be especially prominent in patients with grade C periodontitis and positively correlated with bone loss.

Saliva contains electrolytes such as sodium, potassium, calcium, magnesium, bicarbonate and phosphate. In addition, saliva contains immunoglobulins, proteins, enzymes, mucins and the nitrogenous compounds urea and ammonia. In recent years, saliva has been increasingly recognized as a useful tool in ancillary diagnostic methods. Sialometry and sialochemistry techniques are used in the diagnosis of systemic diseases, in the follow-up of general health status and as a risk indicator for diseases that determine the relationship between oral health and systemic health.

Saliva has been identified as an effective tool for screening and monitoring periodontitis because it is easily collectable and can reflect the inflammatory status of the whole mouth. Indeed, various cytokines and immune mediators present in saliva have been associated with inflammatory processes that progress with unstable responses.

To the best of the author's knowledge, no studies have evaluated salivary GM-CSF and MIP-1α levels in relation to periodontal disease in the existing literature. This study aimed to investigate the changes of these cytokines in the presence of periodontal disease by comparatively examining the levels of GM-CSF, MIP-1α and IL-1β in saliva samples obtained from healthy individuals with gingivitis and periodontitis, to show their potential to be used in the diagnosis of the disease or to provide preliminary information for future treatments that may be performed through these cytokine pathways.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy participants.
* At least twenty permanent teeth present in the oral cavity.
* Non-smokers.
* No medication for continuous use.
* Not pregnant or breastfeeding.

Exclusion Criteria:

* Any oral or systemic disease.
* Regular use of systemic medications.
* Pregnancy or lactation.
* Received periodontal treatment within the last 6 months.
* Use of antibiotics, anti-inflammatory medications, or systemic corticosteroids in the last 6 months.
* Smokers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Systemically healthy, non-smoking adults aged 18-70 years who have not used any medication in the last 6 months, are not pregnant or in the lactation period, and present for routine periodontal examination. Participants are categorized into periodontally healthy, gingivitis, and periodontitis groups based on clinical periodontal parameters
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Salivary level of GM- CSF | 24 hours after taking the clinical measurements at the first visit
  Amount of GM-CSF in human saliva
Salivary level of MIP-1α | 24 hours after taking the clinical measurements at the first visit
  Amount of MIP-1α in human saliva
Salivary level of IL-1β | 24 hours after taking the clinical measurements at the first visit
  Amount of IL-1β in human saliva

SECONDARY OUTCOMES:
Bleeding on Probing | At the initial visit.
  The following index criteria will be used to determine the degree of inflammation in the soft tissue surrounding the vestibular, lingual, mesial and distal surfaces of all teeth. The number of positive (+) scoring areas on the examined surfaces will be calculated as a percentage of the total number of examined areas.
  (-): No bleeding when the periodontal probe is passed along the gingival sulcus.
  (+): Bleeding is present at the gingival margin.
Periodontal Probing Depth | At the initial visit.
  Distance between the gingival margin and sulcus/pocket floor
Clinical Attachment Level | At the initial visit.
  Distance between the enamel-cement junction and the sulcus/base of the pocket.
Plaque Index | At the initial visit.
  For plaque index measurement, values will be obtained from four surfaces of each tooth: mesial, distal, vestibular and palatinal. The values will be summed and divided by four to determine the PI score for each tooth. Scoring will be done as follows; 0: No bacterial plaque on the gingival area of the tooth surface.
  1. No bacterial plaque is visible on the surface of the tooth by eye, but after probing, bacterial plaque is observed at the tip of the probe.
  2. The gingival area is covered with a thin to moderate amount of bacterial plaque, which is visible by eye.
  3. There is a large amount of soft debris, the thickness of which has completely filled the gingival groove and the interdental space is filled with soft debris.
Gingival Index | At the initial visit.
  The vestibule, lingual, mesial and distal surfaces of all teeth will be examined. The values will be summed and divided by four to determine the GI score for each tooth.
  0: Healthy gingiva.
  1. Mild inflammation, mild discoloration and edema but no bleeding after probing.
  2. Moderate inflammation, edema, redness and brightness, bleeding on probing.
  3. Severe inflammation and redness, edema, ulceration and tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Şükrü Enhoş, Prof. Dr., Study Director — Izmir Katip Celebi University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Izmir Katip Çelebi University Department of Periodontology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during the study will not be shared with other researchers or made publicly available. Only summarized results will be disseminated through publications or presentations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available (if applicable) beginning 6 months after publication of the primary results and ending 36 months after publication.
Access Criteria: Qualified researchers with a methodologically sound proposal may request access to the individual participant data (IPD). Proposals should be directed to the Principal Investigator. To gain access, researchers will be required to sign a data access agreement and ensure compliance with ethical data use standards.